CLINICAL TRIAL: NCT06536452
Title: Hematopoiesis in Monoclonal B Cell Lymphocytosis (MBL) and B-Chronic Lymphocytic Leukemia (CLL) Versus Healthy Age-Matched Control Subjects
Brief Title: Hematopoiesis in MBL and CLL Versus Healthy Age-Matched Control Subjects
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 16-006204; NCI-2024-00996 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-006204 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Lymphocytic Leukemia; Monoclonal B-Cell Lymphocytosis
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and bone marrow aspiration and biopsy and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates hematopoiesis to determine how MBL/CLL affected bone marrow responds to fight off infections in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the cellular and mechanistic basis of bone marrow (BM) hematopoietic dysfunction in untreated MBL and CLL patients.

II. Determine if MBL and CLL B cell derived cellular products directly alter the differentiation and functional capacities of Hematopoietic Stem and Progenitor Cells (HSPCs).

III. Utilize the Emu-Tcl1 transgenic mouse model to determine how MBL and CLL patient-derived cellular products alter BM hematopoiesis.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and bone marrow aspiration and biopsy and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects in the CLL cohort who are eligible for these studies will have a clinically established diagnosis of CLL as assessed by flow cytometry and will include subjects who

  * Remain untreated
  * Are currently being treated
  * Who have already been treated
* Subjects in the MBL cohort will have a clinically established diagnosis of MBL
* Healthy age-matched control subjects
* Healthy younger control subjects aged > 40 years

Exclusion Criteria:

* Anyone under 40
* Healthy control subjects must not have a diagnosis of CLL or MBL

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with MBL, patients with CLL ,and healthy subjects recruited through Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-11-18 (Estimated)

PRIMARY OUTCOMES:
Effects of MBL on bone marrow function | Baseline
  Samples collected from healthy participants and participants with MBL will be compared for differences in bone marrow function (i.e., ability to fight off infection). Results will be descriptive. With participant permission, samples will be stored for future research use.
Effects of CLL on bone marrow function | Baseline
  Samples collected from healthy participants and participants with CLL will be compared for differences in bone marrow function (i.e., ability to fight off infection). Results will be descriptive. With participant permission, samples will be stored for future research use.

CONTACTS AND LOCATIONS:
Overall Officials: Neil E. Kay, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials